CLINICAL TRIAL: NCT06214260
Title: Proteomic Profile in Women With Endometriosis (PROTEO-ENDO) Study
Brief Title: Menstrual Blood Proteomic Profile in Women With Endometriosis (PROTEO-ENDO) Study
Acronym: PROTEO-ENDO
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Ronald Wang, Professor & Division head of Obstetrics and Gynaecology, Chinese University of Hong Kong
Other Study IDs: PROTEO-ENDO 20230313
Record Dates: First submitted 2024-01-10; First posted 2024-01-19 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Endometriosis; Endometriosis Ovary; Endometriosis-related Pain
Keywords: Endometriosis; Menstrual blood; Proteomics
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma will be isolated from both peripheral and menstrual blood.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endometriosis: Women suggested endometriosis by clinical presentations & imaging and scheduled for surgical treatment (laparotomy/laparoscopy) at the age of 18-45 years having regular menstrual cycles will be recruited. Finally laparoscopy and histology confirmed endometriosis cases will be eligible for the final analysis.
  Interventions: Diagnostic Test: Peripheral blood sample; Diagnostic Test: Menstrual Blood sample
- Healthy groups: Control subjects at the age of 18-45 years, who have regular menstrual cycles and self-reported no history suggestive of a diagnosis of endometriosis will be recruited.
  Interventions: Diagnostic Test: Peripheral blood sample; Diagnostic Test: Menstrual Blood sample

INTERVENTIONS:
Diagnostic Test: Peripheral blood sample — Peripheral blood will be collected with a 10 ml Ethylenediaminetetra acetic acid (EDTA) tube before surgery during menstrual phase. Additionally, participants will be asked with an interview on demographic, surgical, medical, obstetric, gynecological, contraceptive and medication use history which is validated by Endometriosis Research Foundation Endometriosis Phenome and Biobanking Harmonization Project (WERF EPHect). Pain symptoms before surgery will be evaluated through a 10 cm long one-dimensional visual-analogue scale (VAS).
Diagnostic Test: Menstrual Blood sample — 5ml menstrual blood will be collected before surgery by the women herself. Additionally, participants will be asked with an interview on demographic, surgical, medical, obstetric, gynecological, contraceptive and medication use history which is validated by Endometriosis Research Foundation Endometriosis Phenome and Biobanking Harmonization Project (WERF EPHect). Pain symptoms before surgery will be evaluated through a 10 cm long one-dimensional visual-analogue scale (VAS).

SUMMARY:
In this prospective case control study a total of 66 women (33 women with endometriosis) and (33 healthy women) will be recruited. The main objective of the study is to investigate the proteomic profile of menstrual blood in women with endometriosis compared to controls. Additionally, differentially expressed proteins will be investigated across different stages, clinical presentations, and subtypes of endometriosis

DETAILED DESCRIPTION:
Endometriosis is a disease characterized by the growth of endometrium like tissue outside the uterus. It is the most common and complex gynecological complications in reproductive age woman and schoolgirls. Though the exact etiology of endometriosis is unknown, and the incidence is varying among age and women with infertility, however, it ranges from 2% to 10% within the general female population, estimating around 190 million women at reproductive age and schoolgirls globally and up to 50% in infertile women. The variable, non-specific and broad symptoms of endometriosis lead the clinicians not to easily diagnose the disease and it causes a lengthy delay between the onset of symptoms and confirmation of diagnosis. To date, there is no known non-invasive diagnostic method for endometriosis and no known cure for endometriosis, and treatment is usually aimed at controlling symptoms. New noninvasive non-imaging diagnostic methods, such as biomarkers in serum/blood, and urine have been proposed. However, a definitive diagnosis biomarker is not available yet. Despite the range of blood tests that have been investigated, and altered levels of cancer antigen (CA-125), cytokines, angiogenic, and growth factors, none of the biomarkers showed the definitive diagnosis of endometriosis. Hence this prospective case control study aims to explore non-invasive diagnostic biomarkers from menstrual blood and establish pathophysiology mechanism of the disease. This study is undergoing based on the Helsinki Declaration Guideline for Good Clinical Practice (GCP) standards. Ethical approval is obtained from the Joint Chinese University of Hong Kong and New Territories East Cluster (CUHK-NTEC) Clinical Research Ethics Committee, Hong Kong with reference number: 2023.126.

ELIGIBILITY:
Inclusion Criteria:

* Endometriosis group. are women aged 18-45 years old Laparoscopy with histologically confirmed diagnosis of endometriosis
* Healthy group are women between 18-45 years old self reported no known history of medical & surgical diseases and no any sign of endometriosis related symptoms

Exclusion Criteria:

Endometriosis group

* Hormonal treatment in the past three months before surgery,
* Previous and current malignancy
* Having history of autoimmune disease
* Having previous surgery due to endometriosis
* Pelvic inflammatory disease (PID)
* Lactating/breastfeeding women
* Adenomyosis
* Polycystic ovarian syndrome (PCOS)
* History of or currently on traditional Chinese medicine

  - Healthy group
* Hormonal treatment in the past three months before surgery,
* Previous and current malignancy
* Having history of autoimmune disease
* Having previous surgery due to endometriosis
* Pelvic inflammatory disease (PID)
* Lactating/breastfeeding women
* Adenomyosis
* Polycystic ovarian syndrome (PCOS)
* History of or currently on traditional Chinese medicine

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Given that this study aims to collect menstrual blood and examine differentially expressed proteins, solely individuals of the female gender are deemed eligible
Study Population: Endometriosis group: Patients referred to Obstetrics and Gynaecology specialty outpatient clinic by clinicians for the diagnosis of endometriosis, and/or treatment, or for pelvic pain investigation, and agreed to undergo for laparoscopic surgery for the investigation and/or treatment of endometriosis, or pelvic pain will be recruited.
  Healthy groups: Women who have self-reported that they do not have any known medical, surgical, or gynecological conditions.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2025-11-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Menstrual blood plasma proteomic profile using Liquid chromatography-mass spectrometry (LC-MS/MS) | 24 months
  A functional proteomic assay will be employed to separate a protein to identify the putative novel biomarkers of endometriosis using shotgun proteomics with mass spectrometry. Both expression and functional proteomics will be investigated in women with endometriosis, and controls. A bottom-up proteomics approach will be implemented through steps such as extraction of proteins from a sample, digestion of proteins into peptides, post-digestion separations, and analysis

SECONDARY OUTCOMES:
Determination of menstrual blood plasma proteomic profile in endometriosis phenotypes using an LC-MS/MS | 24 months
  Investigators expect that women in the endometriosis group will differ with regard to proteomic profile with respect to the disease phenotype different phenotypes of the disease: peritoneal endometriosis, ovarian endometriosis, deep infiltrating endometriosis
Menstrual blood plasma proteomic profile in early (stage I/II) and Advance (stage III/IV) stage of endometriosis | 24 months
  According to the revised American society of reproductive medicine (rASRM) endometriosis is categorized in to four stages. The protein expression of each stages of endometriosis will be compared with the bottom-up approach proteomics study using LC-MS/MS
Comparing the plasma of menstrual and peripheral blood proteomic profile using LC-MS/MS | 24 months
  As the composition of menstrual blood is heterogeneous and complex, investigators expect the expressed proteins from the peripheral blood plasma will differ from the expressed proteins of menstrual blood.

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be available as a supplementary file in publications. It will be available to anyone up on the official request from the principal investigator
Supporting Information: Study Protocol, SAP
Time Frame: Two year after initiation of the study
Access Criteria: official request and memorandum of understanding signing